CLINICAL TRIAL: NCT01049412
Title: A Phase 2 Study of LY2605541 Compared With Insulin Glargine in the Treatment of Type 1 Diabetes Mellitus
Brief Title: A Study for Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12151; I2R-MC-BIAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2605541 First, Then Insulin Glargine (Experimental): Participants received LY2605541 for 8 weeks, followed by insulin glargine for 8 weeks.
  Interventions: Drug: LY2605541; Drug: Insulin glargine
- Insulin Glargine First, Then LY2605541 (Active Comparator): Participants received insulin glargine for 8 weeks, followed by LY2605541 for 8 weeks.
  Interventions: Drug: LY2605541; Drug: Insulin glargine

INTERVENTIONS:
Drug: LY2605541 — Administered subcutaneously every morning with dose titration based on blood glucose measures for 8 weeks in each of 2 study periods.
Drug: Insulin glargine — Administered subcutaneously every morning with dose titration based on blood glucose measures for 8 weeks in each of 2 study periods.

SUMMARY:
Comparison of blood glucose levels in patients with Type 1 diabetes when they take a new basal insulin analog and when they take insulin glargine

DETAILED DESCRIPTION:
Prestudy treatment for patients who enter this study will be once daily insulin glargine along with mealtime insulins. Patients will continue to use their mealtime insulins throughout the study. The study will consist of 16 weeks of treatment and 4 weeks of follow-up. The 16 weeks of treatment will consist of two 8-week periods (Periods 1 and 2) during which patients will receive insulin glargine for 8 weeks and LY2605541 for 8 weeks in a random sequence. During the 4-week follow-up period, patients will return to insulin glargine or another basal insulin recommended by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (T1DM) for at least 1 year and using insulin glargine for at least 6 months with a maximum daily dose of 1 unit per kilogram (U/kg).
* Hemoglobin A1c (HbA1c) of no greater than 10.5% before randomization
* Body mass index (BMI) 19 to 45 kilogram per square meter (kg/m²)
* Capable and willing to prepare and inject insulin with a syringe, monitor own blood glucose, complete the study diary, be receptive to diabetes education, comply with study requirements, and receive telephone calls during treatment
* Women of childbearing potential must test negative for pregnancy before receiving treatment and agree to use reliable birth control until completing the follow-up

Exclusion Criteria:

* Twice daily use of insulin glargine within 30 days prior to the study
* Use of any oral or injectable medication intended for the treatment of diabetes mellitus other than insulins in the 3 months prior to the study
* Use of an insulin pump
* More than 1 episode of severe hypoglycemia within 3 months prior to the study, or currently diagnosed as having hypoglycemia unawareness
* 2 or more emergency room visits or hospitalizations due to poor glucose control in the 6 months preceding the study
* Known hypersensitivity or allergy to any of the study insulins or their excipients
* Blood transfusion or severe blood loss within 3 months prior to the study or known hemoglobinopathy, hemolytic anemia, or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the HbA1c methodology
* Irregular sleep/wake cycle
* Pregnant or intend to become pregnant during the study
* Women who are breastfeeding
* Use of prescription or over-the-counter medications to promote weight loss within 3 months prior to the study
* Current participation in a weight loss program or plans to do so during the study
* Use of chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy currently or within 4 weeks prior to the study
* Cardiac disease with a marked impact on physical functioning
* Clinically significant electrocardiogram (ECG) abnormalities at screening
* Fasting triglycerides greater than 500 milligram per deciliter (mg/dL)
* Liver disease
* History of renal transplantation, current renal dialysis, or creatinine greater than 2.0 mg/dL (177 micromole per liter [μmol/L])
* Malignancy other than basal cell or squamous cell skin cancer, currently or within the last 5 years
* Treatment with any antibody-based therapy within 6 months prior to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky

REFERENCES:
- [Background] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287
- [Derived] Rosenstock J, Blevins TC, Bergenstal RM, Morrow LA, Qu Y, Jacober SJ. Reduction in short-acting insulin requirement accompanies improved glycemic control with basal insulin peglispro compared with insulin glargine in patients with type 1 diabetes. J Diabetes. 2016 Jan;8(1):166-9. doi: 10.1111/1753-0407.12332. Epub 2015 Nov 17. No abstract available. PMID 26278063
- [Derived] Rosenstock J, Bergenstal RM, Blevins TC, Morrow LA, Prince MJ, Qu Y, Sinha VP, Howey DC, Jacober SJ. Better glycemic control and weight loss with the novel long-acting basal insulin LY2605541 compared with insulin glargine in type 1 diabetes: a randomized, crossover study. Diabetes Care. 2013 Mar;36(3):522-8. doi: 10.2337/dc12-0067. Epub 2012 Nov 27. PMID 23193209

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label, randomized, 2-arm crossover study. The study consisted of two 8-week periods (Periods I and II) during which participants received Glargine for 8 weeks and LY2605541 for 8 weeks in a random sequence.
Groups:
- LY2605541/Glargine: Participants took LY2605541 in Period I and Glargine in Period II
- Glargine/LY2605541: Participants took Glargine in Period I and LY2605541 in Period II
Period: Period I
Arm/Group | LY2605541/Glargine | Glargine/LY2605541
Started | 70 | 68
Took at Least One Dose of Study Drug | 69 | 68
Completed | 62 | 55
Not Completed | 8 | 13
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Adverse Event | 1 | 0
Period: Period II
Arm/Group | LY2605541/Glargine | Glargine/LY2605541
Started | 62 | 55
Completed | 58 | 52
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2605541/Glargine | Glargine/LY2605541 | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.82 (11.34) | 39.53 (12.28) | 38.17 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 41 | 45 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  Multiple | 1 | 0 | 1
  White | 65 | 64 | 129
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 64 | 126
  Israel | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Daily Average Blood Glucose (Avg. BG) at Week 8 Endpoint as Measured by the 8-Point Self-Monitored Blood Glucose (SMBG) Profiles
Description: It is the Avg. of the 8-point SMBG profiles, BG of morning fasting, midday & evening pre-meal, 2-hour postprandial after each of the 3 main meals, bedtime, 0300 hours. Least squares (LS) mean of daily Avg. BG is from mixed-model repeated measures (MMRM), which includes fixed effects of treatment (LY2605541, Glargine); Treatment Sequence; treatment period; dose conversion (pre-interim analysis [IA], post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline Hemoglobin [HbA1c] group); visit; visit and treatment interaction; a random effect for participant.
Time Frame: Week 8 of each treatment period
Population: All randomized participants who took at least one dose of study drug with non-missing baseline value and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: millimole per Liter (mmol/L)
Groups:
- Glargine: Administered subcutaneously every morning with dose titration based on blood glucose measures for 8 weeks in each of 2 study periods
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 92 | 91
millimole per Liter (mmol/L) | 7.98 (0.32) | 8.53 (0.33)
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = -0.55, 90% CI 2-sided [-0.81 to -0.29], Standard Error of Mean 0.16

2. Secondary Outcome: Change From Baseline in Daily Average Blood Glucose (Avg. BG) at Week 8 Endpoint as Measured by the 8-Point Self-Monitored Blood Glucose (SMBG) Profiles
Description: It is the Avg. of the 8-point SMBG profiles, BG of morning fasting, midday & evening pre-meal, 2-hour postprandial after each of the 3 main meals, bedtime, 0300 hours. LS mean of daily Avg. BG is from MMRM, which includes fixed effects of treatment (LY2605541, Glargine); Treatment Sequence; treatment period; dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; a random effect for participant.
Time Frame: Baseline, Week 8 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 92 | 91
mmol/L | -0.74 (0.40) | -0.18 (0.40)
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = -0.56, 90% CI 2-sided [-0.83 to -0.29], Standard Error of Mean 0.16

3. Secondary Outcome: Change From Baseline in Hemoglobin (HbA1c) at Week 8 Endpoint of Period I
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean of the change from baseline to 8-week at Period I is from MMRM approach, which includes fixed effects of treatment (LY2605541, Glargine); dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group); baseline HbA1c; visit; interaction between visit and treatment; and a random effect for participant.
Time Frame: Baseline, Week 8 (Period I)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 62 | 54
percentage of glycated hemoglobin | -0.45 (0.10) | -0.34 (0.11)
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.242, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = -0.11, 90% CI 2-sided [-0.28 to 0.05], Standard Error of Mean 0.10

4. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and HbA1c ≤6.5% at Week 8 Endpoint of Period I
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 8 (Period I)
Population: All randomized participants who took at least one dose of study drug with non-missing baseline value and at least one non-missing post-baseline value, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 65 | 60
percentage of participants
  HbA1c <7.0% | 43.1 | 33.3
  HbA1c ≤6.5% | 24.6 | 13.3
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.276, Fisher Exact — The statistical significance level is 0.10. P-value is for HbA1c <7.0%
Statistical Analysis 2: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.119, Fisher Exact — The statistical significance level is 0.10. P-value is for HbA1c ≤6.5%

5. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and HbA1c ≤6.5% at Week 8 Endpoint Who Did Not Experience a Hypoglycemic Episode During Treatment (Period I)
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 millimole/Liter (mmol/L) (≤70 milligram/deciliter [mg/dL]) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005]).
Time Frame: Week 8 (Period I)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 65 | 60
percentage of participants
  HbA1c <7.0% | 1.5 | 1.7
  HbA1c ≤6.5% | 0 | 0

6. Secondary Outcome: 8-Point Self-Monitored Blood Glucose (SMBG) Measures at Week 8 Endpoint
Description: 8-point SMBG profiles are measured at morning fasting BG (FBG), midday pre-meal BG, evening pre-meal BG, 2-hour postprandial BG after each of the 3 main meals, bedtime BG, 0300 hours BG. LS mean is obtained from MMRM approach, which includes fixed effects of treatment (LY2605541, Glargine); treatment sequence; treatment period; dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; interaction between visit and treatment; and a random effect for participant.
Time Frame: Week 8 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 124 | 130
mmol/L
  0300 hours BG: number analyzed (Participants) | 98 | 94
  0300 hours BG | 8.97 (0.50) | 8.67 (0.51)
  Morning FBG: number analyzed (Participants) | 105 | 102
  Morning FBG | 9.33 (0.45) | 9.57 (0.49)
  Morning 2-hr postprandial BG: number analyzed (Participants) | 103 | 102
  Morning 2-hr postprandial BG | 8.27 (0.46) | 8.76 (0.46)
  Midday Pre-meal BG: number analyzed (Participants) | 105 | 102
  Midday Pre-meal BG | 6.98 (0.43) | 7.52 (0.45)
  Midday 2-hr postprandial BG: number analyzed (Participants) | 105 | 101
  Midday 2-hr postprandial BG | 8.08 (0.44) | 8.60 (0.47)
  Evening Pre-meal BG: number analyzed (Participants) | 104 | 102
  Evening Pre-meal BG | 7.87 (0.38) | 8.73 (0.41)
  Evening 2-hr postprandial BG: number analyzed (Participants) | 105 | 102
  Evening 2-hr postprandial BG | 8.37 (0.44) | 9.26 (0.46)
  Bed time BG: number analyzed (Participants) | 101 | 99
  Bed time BG | 8.20 (0.45) | 9.29 (0.48)
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.392, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for 0300 hour BG; Least Squares Mean Difference (Final) = 0.30, 90% CI 2-sided [-0.28 to 0.88], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.464, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for morning FBG; Least Squares Mean Difference (Final) = -0.24, 90% CI 2-sided [-0.79 to 0.30], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.151, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for morning 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.48, 90% CI 2-sided [-1.04 to 0.07], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for midday pre-meal BG; Least Squares Mean Difference (Final) = -0.54, 90% CI 2-sided [-1.05 to -0.03], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.070, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for midday 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.52, 90% CI 2-sided [-0.99 to -0.05], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for evening pre-meal BG; Least Squares Mean Difference (Final) = -0.86, 90% CI 2-sided [-1.39 to -0.34], Standard Error of Mean 0.32
Statistical Analysis 7: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for evening 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.89, 90% CI 2-sided [-1.38 to -0.41], Standard Error of Mean 0.29
Statistical Analysis 8: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for bed time BG; Least Squares Mean Difference (Final) = -1.10, 90% CI 2-sided [-1.64 to -0.55], Standard Error of Mean 0.33

7. Secondary Outcome: Daily Basal Insulin Dose at Week 2 and Week 8 Endpoint
Description: LS mean is obtained from MMRM approach, which includes fixed effects of treatment (LY2605541, Glargine); treatment sequence; treatment period; dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; interaction between visit and treatment; and a random effect for participant.
Time Frame: Week 2 and Week 8 of each treatment period
Population: All randomized participants who took at least one dose of study drug with at least one non-missing value of the response variable at any of the subsequent weeks.
Measure: Least Squares Mean (Standard Deviation); unit: nanomoles per kilogram (nmoles/kg)
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 124 | 130
nanomoles per kilogram (nmoles/kg)
  Week 2: number analyzed (Participants) | 120 | 121
  Week 2 | 3.35 (0.16) | 2.58 (0.16)
  Week 8: number analyzed (Participants) | 116 | 115
  Week 8 | 4.12 (0.18) | 2.86 (0.16)

8. Secondary Outcome: Pharmacokinetics - Drug (LY2605541) Concentration at Steady State (Css) at Week 8 Endpoint
Description: The drug (LY2605541) concentration at steady state (Css) is calculated from the clearance (Liter/hour) and the final dose of the participants. Clearance was estimated using population-based approaches.
Time Frame: Week 8 of each treatment period
Population: Participants who took at least one dose of study drug and had measurements at Week 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per liter (pMol/L)
Arm/Group | LY2605541
Number analyzed (Participants) | 115
picomoles per liter (pMol/L) | 2873 (54.9)

9. Secondary Outcome: Percentage of Participants With Antibody Status Change From Baseline to Week 8, Week 16 and Week 20
Description: Negative is defined as either 'negative' from lab or percent binding <1.16%. Positive is defined as the percent binding is ≥1.16%. The antibody status change is from negative to positive or positive to negative.
Time Frame: Week 8, Week 16 and Week 20
Population: All randomized participants who took at least one dose of study drug with both baseline and endpoint antibody measurements.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541/Glargine | Glargine/LY2605541
Number analyzed (Participants) | 69 | 68
percentage of participants
  Week 8 (Period I) from negative to positive | 8.3 | 3.3
  Week 8 (Period I) from positive to negative | 3.3 | 5.0
  Week 16 (Period II) from negative to positive | 12.5 | 7.4
  Week 16 (Period II) from positive to negative | 1.8 | 7.4
  Week 20 (follow up) from negative to positive | 14.8 | 11.5
  Week 20 (follow up) from positive to negative | 1.9 | 3.8

10. Secondary Outcome: Percentage of Participants With Hypoglycemia Baseline Through Week 8
Description: Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 millimole per Liter (mmol/L) (≤70 milligram per deciliter [mg/dL]) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005].
Time Frame: Baseline through Week 8 of each treatment period
Population: All randomized participants who took at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 124 | 130
percentage of participants | 92.7 | 90.0

11. Secondary Outcome: Rate of Hypoglycemia Per 30 Days Baseline Through Week 8
Description: Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 mmol/L (≤70 mg/dL) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005]. Hypoglycemia rate per 30 days is calculated as the number of hypoglycemia/number of days at risk*30.
Time Frame: Baseline through Week 8 of each treatment period
Population: All randomized participants who took at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: number of hypoglycemia episodes/30 days
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 124 | 130
number of hypoglycemia episodes/30 days | 8.74 (7.70) | 7.36 (6.80)
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p = 0.037, Negative Binomial Model — The statistical significance level is 0.10

12. Secondary Outcome: Glycemic Variability in Fasting Blood Glucose (FBG) at Week 8 Endpoint
Description: Within-patient glycemic variability was assessed as the standard deviation of fasting blood glucose each day between Week 6 and Week 8. LS mean is obtained from MMRM approach, which includes fixed effects of treatment (LY2605541, Glargine); treatment sequence; treatment period; dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; interaction between visit and treatment; and a random effect for participant.
Time Frame: Week 8 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 107 | 107
mmol/L | 3.13 (0.23) | 3.60 (0.24)
Statistical Analysis 1: Comparison: LY2605541 vs Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = -0.47, 90% CI 2-sided [-0.69 to -0.25], Standard Error of Mean 0.13

ADVERSE EVENTS:
Groups:
- LY2605541: Participants took LY2605541 administered subcutaneously every morning with dose titration based on blood glucose measures for 8 weeks
- Glargine: Participants took Glargine administered subcutaneously every morning with dose titration based on blood glucose measures for 8 weeks
Arm/Group | LY2605541 | Glargine
Serious Adverse Events (participants affected / at risk) | 6/125 | 4/130
Other Adverse Events (participants affected / at risk) | 66/125 | 59/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (N=125) | Glargine (N=130)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Severe hypoglycaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (N=125) | Glargine (N=130)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Onychomycosis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 7 (7)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days